CLINICAL TRIAL: NCT04284267
Title: Neuromodulation for Enhancement of Emotion Regulation in Bipolar Mood Disorders
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Kristen K. Ellard, Ph.D., Director of Dimensional Neuroimaging Research, Massachusetts General Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2020P000120
Record Dates: First submitted 2020-02-20; First posted 2020-02-25 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Bipolar Disorder
Keywords: Transcranial Magnetic Stimulation; Emotion Regulation
MeSH Terms: conditions — Bipolar Disorder; Emotional Regulation | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: There will be a healthy control group and a bipolar disorder group. The bipolar disorder group will then be randomized to one of three conditions.
Who Masked: Participant
Masking Description: Masking will be implemented using a active-placebo TMS coil.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Healthy Control (No Intervention): This group consists of individuals with no psychiatric diagnosis.
- Bipolar Group (Experimental): This group consists of individuals with a diagnosis of bipolar disorder who have been randomized to receive high-dose TMS (i.e., 1800 pulses) and sham TMS.
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — TMS is a non-invasive tool for modulating patterns of brain activation and circuit connectivity. It uses electromagnetic pulses to induce electric currents over the cortex that serve to depolarize or hyperpolarize neurons, thereby changing patterns of synaptic activity. This study will use intermittent theta burst stimulation (iTBS), an efficient TMS protocol that uses high frequency (50Hz) triplets of TMS given every 200 milliseconds (i.e. at 5 Hz).
  Other Names: TMS
  Arms: Bipolar Group

SUMMARY:
The investigators are conducting this research study to better understand how individuals with bipolar disorder regulate their emotions, and if transcranial magnetic stimulation (TMS) can help improve emotion regulation for individuals with bipolar mood disorders.

DETAILED DESCRIPTION:
The objective of this study protocol is to test whether intermittent theta-burst transcranial magnetic stimulation (iTBS-TMS) to ventrolateral prefrontal cortex (VLPFC) or inferior parietal lobule (IPL) can improve performance on emotion regulation tasks in patients with bipolar disorder. Results from this study will help inform future treatment development to improve emotion regulation in patients with bipolar disorder. The study will proceed in two phases: During Phase 1, a cohort of 30 healthy control subjects will be recruited in order to establish a normative sample from which to compare patient data. Functional magnetic resonance imaging (fMRI) data will be collected from healthy control participants during performance on two emotion regulation tasks (probing implicit and explicit emotion regulation). Data from these subjects will provide a normative distribution of VLPFC and IPL function from which to compare individual patients. During Phase 2, a cohort of 30 patients diagnosed with bipolar disorder will be recruited. Patient participants will perform the same two emotion regulation tasks during fMRI scanning. Data from individual patients will be analyzed to detect specific VLPFC and IPL subregions showing activation deviations from healthy controls (Phase 1 data). Patient-specific VLPFC and IPL subregions showing patterns of activation greater than two standard deviations from healthy controls will be used as individualized target sites for TMS stimulation. Patients will then receive high-dose iTBS-TMS (1800 pulses) of the VLPFC and IPL, and sham iTBS-TMS to the dorsomedial prefrontal cortex (dmPFC) across three separate study visits. Order of target stimulation will be randomized across participants. TMS sessions will take approximately 10 minutes and will be immediately followed by an fMRI scanning session, during which participants will again complete the implicit and explicit emotion regulation tasks. TMS sessions will take place in the scanning bay to enable quick transition to the fMRI task. Baseline scanning sessions and either active TMS-fMRI or sham TMS-fMRI sessions will occur on separate days, no more than two weeks apart. Effects of iTBS-TMS on emotion regulation will be evaluated by comparing pre-TMS versus post-TMS behavior, neural activation, and functional connectivity patterns during performance on implicit and explicit emotion regulation tasks.

ELIGIBILITY:
Inclusion Criteria (Healthy Controls)

1. Male or female age 18-55
2. No history of psychiatric disorder, as assessed using the Mini-International Neuropsychiatric Interview (MINI).
3. Non-Clinical Levels of Emotion Dysregulation, as assessed using the Difficulties in Emotion Regulation Scale (DERS) Non-clinical levels of emotion dysregulation will be defined as a score < 80 on the DERS.

Exclusion Criteria (Healthy Controls)

1. Current or history of psychiatric disorders
2. Endorsement of clinical levels of emotion dysregulation
3. Current or history of: organic mental disorder; substance abuse within the past 12 months and/or history of substance abuse for > 1 year; past or current substance dependence (including alcohol); schizophrenia; delusional disorder; and psychotic disorders.
4. Current pregnancy.
5. Medical illness or non-psychiatric medical treatment that would likely interfere with study participation
6. Neurologic disorder, prior neurosurgical procedure, prior electroconvulsive therapy (ECT) or TMS, history of seizures or head trauma.
7. Presence of metallic implants that would interfere with safety during fMRI scanning.

Inclusion Criteria (Bipolar Disorder Group)

1. Male or female age 18-55
2. Diagnosis of Bipolar I Disorder (BD-I), as assessed through MINI.
3. Current mood state euthymic.

   a. Hamilton-Depression Rating Scale (HAM-D-17) and Young Mania Rating Scale (YMRS) will be used to assess current depressive and manic symptoms. Euthymia will be defined as a HAM-D-17 score <10 and YMRS score <12.
4. Clinical Levels of Emotion Dysregulation, as assessed using the DERS. Clinical levels of emotion dysregulation will be defined as a score > 80 on the DERS.

Exclusion Criteria (Bipolar Disorder Group)

1. Current symptoms of mania or depression (YMRS score >12, HAM-D-17 score >10).
2. Medication instability (<3 months).
3. Current or history of: organic mental disorder; substance abuse within the past 12 months and/or history of substance abuse for > 1 year; past or current substance dependence (including alcohol), verified by urine toxicology screen; schizophrenia; delusional disorder; and psychotic disorders.
4. Current pregnancy.
5. Medical illness or non-psychiatric medical treatment that would likely interfere with study participation
6. Neurologic disorder, prior neurosurgical procedure, prior ECT or TMS, history of seizures or head trauma.
7. Presence of metallic implants that would interfere with safety during fMRI scanning.

Ages: 22 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Multisource Interference Task with International Affective Pictures Set (MSIT-IAPS) | Change from Baseline to Post-TMS Stimulation (30 min-1 hour)
  The MSIT-IAPS task is a well-validated fMRI task designed to assess the effects of emotional distractors on cognitive control. During each trial, a three-digit number is presented. Each set contains two identical distractor numbers and a target number that differed from the distractors. Participants report via a button press the identity of the target number that differs from the two distractor numbers. Noninterference (control) trials: distractor numbers are always zeros, and the identity of the target number always corresponds to its position on the button response pad (100, 020, 003). Interference trials: distractor numbers are always numbers other than 0, and the identity of the target number is always incongruent with its position on the button response pad (e.g. 211, 232, 331, etc.). Each trial of the MSIT is overlaid on a negative, positive, or neutral IAPS image. Reaction time (ms) and accuracy (% correct) is calculated for each trial.
Emotion Conflict Resolution Task | Change from Baseline to Post-TMS Stimulation (30 min-1 hour)
  The ECR task is a well-validated task designed to assess the effects of emotional conflict that arises from the incompatibility between task-relevant and task-irrelevant emotional dimensions of a stimulus. Faces with fearful and happy expressions are presented with the words "happy" or "fear" written across them. Words are either congruent (e.g. "happy" written across an image with a happy expression) or incongruent (e.g. "happy" written across an image with a fearful expression). Subjects are asked to identify the emotional expression of the face while ignoring the word. Trials are analyzed with regard to immediately preceding trials: incongruent trials preceded by congruent trials (CI trials) measure emotion conflict, and incongruent trials preceded by incongruent trials (II trials) measure resolution of emotion conflict. Reaction time (ms) and accuracy (% correct) is calculated for each trial.

SECONDARY OUTCOMES:
MSIT-IAPS Task-induced blood oxygen level dependent (BOLD) signal | Change from Baseline to Post-TMS Stimulation (30 min-1 hour)
  Task-dependent linear time course (ß-value) of BOLD signal during performance of MSIT-IAPS task. Differences in ß-values during relevant task conditions (CI versus II) are compared.
MSIT-IAPS Task-induced blood oxygen level dependent (BOLD) signal functional connectivity | Change from Baseline to Post-TMS Stimulation (30 min-1 hour)
  Task-dependent BOLD signal correlation strengths (z-transformed values) during performance of the task. Differences in z-transformed values during relevant task conditions (CI versus II) are compared.
ECR Task-induced blood oxygen level dependent (BOLD) signal | Change from Baseline to Post-TMS Stimulation (30 min-1 hour)
  Task-dependent linear time course (ß-value) of BOLD signal during performance of the Cognitive Reappraisal task. Differences in ß-values during relevant task conditions (Reappraise versus Attend) are compared.
ECR Task-induced blood oxygen level dependent (BOLD) signal functional connectivity | Change from Baseline to Post-TMS Stimulation (30 min-1 hour)
  Task-dependent BOLD signal correlation strengths (z-transformed values) during performance of the Cognitive Reappraisal task. Differences in ztransformed values during relevant task conditions (Reappraise versus Attend) are compared.
Skin Conductance Response | Change from Baseline to Post-TMS Stimulation (30 min-1 hour)
  Skin conductance response is measured by recording electrodermal skin response using electrode sensors applied to fingertips. Correlation between changes in skin conductance response and changes in task performance (RT, distress ratings) are examined as a task manipulation check.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Ellard, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Martinos Center for Biomedical Imaging, Charlestown, Massachusetts, United States